CLINICAL TRIAL: NCT01331369
Title: Intensification of Care to Improve Adherence to Anti-hypertensives in Primary Care: a Pragmatic Clinical Trial.
Brief Title: Intensification of Care to Improve Adherence to Anti-hypertensives
Acronym: HyperCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade de Blumenau (Other)
Collaborators: Fundacao de Apoio a Pesquisa de Santa Catarina (Unknown)
Responsible Party: Principal Investigator, Ernani Tiaraju de Santa Helena, Professor, Universidade de Blumenau
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FURB 2010/01
Record Dates: First submitted 2011-03-29; First posted 2011-04-08 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Medication Adherence
Keywords: adherence; compliance; persistence; drop out; abandon
MeSH Terms: conditions — Medication Adherence; Patient Compliance | interventions — Comprehensive Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Usual care. It means routine medical care that include free demand consultation and free medicines.
  Interventions: Other: Usual Care
- Intervention (Experimental): Intensification of care. Besides routine medical care that include free demand consultation and free medicines, subjects were invited to have 6 structured medical encounters based on a social-psychological approach. Doctors must follow a protocol to conduct the encounter that have around 30 minutes each.
  Interventions: Behavioral: Intensification of Care

INTERVENTIONS:
Behavioral: Intensification of Care — Usual provided care plus social-psychological intervention: 6 consultation with doctors and 9 with community health workers, both oriented by protocol.
  Other Names: Comprehensive Care
  Arms: Intervention
Other: Usual Care — Usual care provided (medical and/or nurse consultation and medicines)
  Other Names: Usual
  Arms: Control

SUMMARY:
The aim of the study is to evaluate the effectiveness of a social-psychological intervention to improve anti-hypertensives adherence in primary care. Its is a pragmatic clinical trial.

DETAILED DESCRIPTION:
We will study two groups of 198 people with hypertension treated in ten health care units. One group will receive usual care dispensed in units (control). The other group (intervention) will be offered six individual assistance with health care worker physician or nurse) during the period of 9 months with a minimum interval of 30 days, plus 9 monthly visits structured by community health agents. Adherence will be measured in both groups at baseline and months 3, 6, 9 and 12, through validated questionnaire and pill count. Also evaluated clinical outcome measures (blood pressure, hospitalizations and deaths). The analysis will be done by intention to treat comparing adherence measures and clinical outcome between groups (Student t test and chi-square test) and within groups over time (paired t test and McNemar). It will be accepted p value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* persons with hypertension aged 18 years and older

Exclusion Criteria:

* those with physical or mental impaired that cannot go to health care units or cannot answer a questionnaire
* pregnants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of people adherent to treatment - MMAS-8 | at basal and 3, 6, 9 and 12 months
  It will be measure by "Moriski Medication Adherence Scale 8 item", translated and validated in Brazil. MMAS scores were trichotomized previously into the following 3 levels of adherence: high adherence (score, 8), medium adherence (score, 6 to <8), and low adherence (score, <6).

SECONDARY OUTCOMES:
Change in the proportion of people adherent to treatment - QAM-Q | at basal and 3, 6, 9 and 12 months
  It will be measure by "Questionário de Adesão a Medicamentos -Qualiaids" 3 item, an structured questionnaire developed and validated in Brazil. Non-adherence was accepted if respondent doesn't take 80% of his medicines or if he/she presents any errors on the process (time, jumps..)
Means difference and/or risk ratio between and within groups of clinical outcomes | at basal and 3, 6, 9 and 12 months
  It will be evaluated mean blood pressure, proportion of complications, hospitalization and death in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Ernani S Helena, PhD, Principal Investigator — Regional University of Blumenau
Locations (1):
- Family Health Units - Unique Health System, Blumenau, Santa Catarina, Brazil

REFERENCES:
- See also: Research Group of Pharmacoepidemiology — http://dgp.cnpq.br/dgp/espelhogrupo/4971570719283133